CLINICAL TRIAL: NCT00816439
Title: Imaging Cannabinoid CB1 Receptors in Alcohol Dependence
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090040; 09-M-0040
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2014-08-28

CONDITIONS: Alcoholism
Keywords: Positron Emission Tomography; Brain Imaging; Alcoholism
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The cannabinoid type 1 (CB1) receptor is a protein found in the brain that is involved with the effects of marijuana; it may also play a role in the effects of alcohol dependence and withdrawal. Earlier animal studies have shown that although long-term alcohol use decreases the number of CB1 receptors in the brain, the number returns to normal after alcohol use stops. This study will use positron emission tomography (PET) and magnetic resonance imaging (MRI) scans to trace a radioactive chemical called [11C]MePPEP, which can locate and measure the number of CB1 receptors in the brain. Researchers will study the CB1 receptors in the brains of people with alcohol dependence, and compare the results to the CB1 receptors in the brains of people without alcohol dependence. The results of this study will be used to further research into appropriate treatment procedures for alcohol dependence.

This study will include 30 men with alcohol dependence and 50 men without alcohol dependence. All of the men must be between 18 and 65 years of age. Participants in both groups must not have any medical conditions that will prevent them from undergoing PET or MRI scans.

For the PET scan, participants will be injected with a small amount of [11C]MePPEP and will then be brought to the PET scanner. The scan will take between 3 and 4 hours, but participants will be allowed to take breaks over the course of the scan. The MRI scan will not require any injections and will take approximately 1 hour to complete.

Participants without alcohol dependence will make three visits to the National Institutes of Health Clinical Center. Blood and urine samples will be taken during one visit, and participants will arrange to have an MRI scan on one visit and a PET scan on the other visit, in whichever order they prefer.

Participants with alcohol dependence will undergo two PET scans: the first will be performed between 3 and 7 days after the participant last consumed alcohol, and the second will be performed approximately 2 to 4 weeks after the first scan (with no alcohol consumption permitted in the interval). Participants will alcohol dependence will also undergo an MRI scan and will provide blood and urine samples.

DETAILED DESCRIPTION:
Alcohol dependence (alcoholism) is a chronic medical illness with a relapsing course and a major public health problem. Alcoholism is clinically characterized by periods of uncontrolled alcohol consumption and withdrawal, during which counter-adaptive mechanisms such as stress and dysphoria are recruited. Neurobiological research into the pathophysiology of the illness suggest that both the primary rewarding effects of ethanol as well as neuroadaptive changes that occur during chronic alcohol exposure involve persistent changes in various brain neurotransmission systems, such as the dopamine, glutamate, and gamma-amino butyric acid (GABA) systems. Recent views of the illness also emphasize the long-lasting recruitment of the brain stress system. Unfortunately, despite this progress, available pharmacological agents for the treatment of alcoholism are too few and not sufficiently efficacious.

The brain endocannabinoid (EC) system is a recently discovered brain neurotransmission system, which involves endogenous cannabinoid agents (ECs) that act upon specific receptors (CB1 and CB2). CB1 receptor is abundant in the human brain and acts as an inhibitory modulator of classical neurotransmitters. ECs and CB1 receptors appear to modulate the brain reward system, and animal studies have demonstrated an important role of CB1 receptor stimulation in alcohol- and drug-related behaviors. During chronic alcohol exposure, EC levels in the brain are elevated and CB1 receptor levels are consequently reduced; this appears to be reversible following withdrawal. Animal studies suggest that CB1 receptor blockade in the abstinent phase may reduce alcohol craving and relapse. To what extent ECs and CB1 receptors are involved in the pathophysiology of alcohol dependence in humans is currently unknown. The lack of suitable methods to reliably quantify CB1 receptors in the living human brain has to date hindered the progress in this field.

In this protocol, we outline studies aiming at elucidating the role of CB1 receptors in alcohol and cannabis dependence by using positron emission tomography (PET) and the recently developed radiotracer for CB1 receptors, [(18)F]FMPEP-d2. The aim of this project is to explore CB1 receptor abnormalities at various stages of alcohol and cannabis dependence in humans. For the studies in alcohol dependence, the primary hypothesis is that CB1 receptors are downregulated during chronic alcohol exposure and upregulated during extended abstinence. For the studies in cannabis users, our primary hypothesis is that CB1 receptors are downregulated during chronic cannabis use and upregulated during extended abstinence. Insight into the role of CB1 receptor function in human alcoholism and in chronic cannabis use may help guide future development of pharmacotherapies.

ELIGIBILITY:
* INCLUSION CRITERIA:

ALCOHOL DEPENDENT SUBJECTS:

1. All subjects must be male, 18-65 years of age and be able to give written informed consent.
2. All subjects must be healthy based on history and physical examination.
3. Subjects must fulfill DSM-IV criteria (American Psychiatric Association 1987) for alcohol dependence. In addition, they must have an alcohol consumption of 35 or more standard drinks per week, as measured by timeline follow-back during the 28-day period preceding admission, as well as during the 7-day period immediately preceding it.
4. About half of the patients with alcohol dependence will be carriers of the C allele of the rs2023239 SNP and half will not.

HEALTHY SUBJECTS:

1. All subjects must be male, 18-65 years of age and be able to give written informed consent.
2. This comparison group must be healthy based on history and physical examination.
3. About half of the healthy subjects will currently smoke cigarettes and about half will not.
4. About half of the healthy subjects will be carriers of the C allele of the rs2023239 SNP and half will not.

CANNABIS USERS:

1. All subjects must be male, 18-65 years of age and be able to give written informed consent.
2. All subjects must be healthy based on history and physical examination.
3. Self-reported cannabis use of at least one year with a typical pattern of use of at least 5 days per week for the six months prior to unit admission.
4. A positive urine cannabinoid test within 90 days of admission.

EXCLUSION CRITERIA:

ALCOHOL DEPENDENT PATIENTS:

1. Any serious medical condition as judged by the investigator in consultation with the attending physician in the NIAAA program.
2. Clinically significant coagulopathies or laboratory abnormalities other than those related to alcohol dependence.

Past or present diagnosis of schizophrenia, bipolar illness or any other psychotic disorder; any current disorder that has required psychoactive medication (other than oxazepam) within the preceding 28-day period (42 days for fluoxetine). 3. Oxazepam is a relatively short acting benzodiazepine and is used clinically during alcohol withdrawal. Any present substance abuse other than alcohol.

4. Positive test for HIV.

5. Metallic foreign bodies that would be affected by the MRI scanner magnet, or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan.

6. Head trauma resulting in a period of unconsciousness lasting longer than 1 hour.

7. History of fetal alcohol syndrome or other neurodevelopmental disorder.

8. History of seizures, other than in childhood and related to fever.

9. Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.

10. Positive urine drug screen.

11. Inability to lie flat on camera bed for about 2.5 h

HEALTHY SUBJECTS:

1. Any current Axis I diagnosis; and any lifetime diagnosis of drug abuse or dependence.
2. Clinically significant laboratory abnormalities.
3. Recent heavy use of alcohol. That is, subjects must have an alcohol audit score of less than or equal to 9. In addition, subjects must agree not to consume any alcohol in the three days prior to the PET scan.
4. Psychotropic medication use (including benzodiazepines and illicit drugs) during the 28 days (42 day for fluoxetine) prior to the PET scan.
5. Serious medical problems.
6. Positive test for HIV.
7. Metallic foreign bodies that would be affected by the MRI magnet, or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan.
8. Head trauma resulting in a period of unconsciousness lasting longer than 10 minutes.
9. History of fetal alcohol syndrome or other neurodevelopmental disorder.
10. History of seizures, other than in childhood and related to fever.
11. Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.
12. Positive urine drug screen.
13. Inability to lie flat on camera bed for about 2.5 h

EXCLUSION CRITERIA: CANNABIS USERS:

1. History or presence of any clinically significant illness, as determined by history, physical examination, and/or laboratory tests.
2. Past or present diagnosis of schizophrenia, bipolar illness or any other psychotic disorder; any current disorder that has required psychoactive medication within the preceding 28-day period (42 days for fluoxetine).
3. Current physical dependence on any substance other than cannabis, nicotine, or caffeine;
4. Positive test for HIV.
5. Metallic foreign bodies that would be affected by the MRI scanner magnet, or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan.
6. Head trauma resulting in a period of unconsciousness lasting longer than 10 minutes.
7. History of fetal alcohol syndrome or other neurodevelopmental disorder.
8. History of seizures, other than in childhood and related to fever.
9. Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.
10. Inability to lie flat on camera bed for about 2.5 h.
11. Regular use of alcohol (greater than or equal to 6 standard drinks per day) four or more times per week in the month prior to study entry.
12. Currently interested in or participating in drug abuse treatment, or participated in drug abuse treatment within 60 days preceding study enrollment.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-12-29; Study Completion 2014-08-28

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Basavarajappa BS, Hungund BL. Role of the endocannabinoid system in the development of tolerance to alcohol. Alcohol Alcohol. 2005 Jan-Feb;40(1):15-24. doi: 10.1093/alcalc/agh111. Epub 2004 Nov 18. PMID 15550443
- [Background] Brown AK, George DT, Fujita M, Liow JS, Ichise M, Hibbeln J, Ghose S, Sangare J, Hommer D, Innis RB. PET [11C]DASB imaging of serotonin transporters in patients with alcoholism. Alcohol Clin Exp Res. 2007 Jan;31(1):28-32. doi: 10.1111/j.1530-0277.2006.00261.x. PMID 17207098
- [Background] Cippitelli A, Bilbao A, Hansson AC, del Arco I, Sommer W, Heilig M, Massi M, Bermudez-Silva FJ, Navarro M, Ciccocioppo R, de Fonseca FR; European TARGALC Consortium. Cannabinoid CB1 receptor antagonism reduces conditioned reinstatement of ethanol-seeking behavior in rats. Eur J Neurosci. 2005 Apr;21(8):2243-51. doi: 10.1111/j.1460-9568.2005.04056.x. PMID 15869521
- [Derived] Hirvonen J, Zanotti-Fregonara P, Gorelick DA, Lyoo CH, Rallis-Frutos D, Morse C, Zoghbi SS, Pike VW, Volkow ND, Huestis MA, Innis RB. Decreased Cannabinoid CB1 Receptors in Male Tobacco Smokers Examined With Positron Emission Tomography. Biol Psychiatry. 2018 Nov 15;84(10):715-721. doi: 10.1016/j.biopsych.2018.07.009. Epub 2018 Jul 21. PMID 30121138